CLINICAL TRIAL: NCT02224027
Title: Comparison of Proceal Laryngeal Mask Airway and I-gel to Machintoch Laryngoscope by Novice Operators in Simulated Difficult Airway - a Manikin Study.
Brief Title: Comparison of Laryngeal Mask and I-gel to Laryngoscope by Novice Operators in Simulated Difficult Airway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sangjin Park, assistant professor, Yeungnam University College of Medicine
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: apsj0821
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- i-gel (Active Comparator): Each novice performs i-gel insertion in difficult laryngoscopy scenario.
  Interventions: Device: i-gel
- proceal laryngeal mask airway (Active Comparator): Each novice performs proceal laryngeal mask airway insertion in difficult laryngoscopy scenario.
  Interventions: Device: proceal laryngeal mask airway
- tracheal tube (Active Comparator): Each novice performs tracheal intubation in difficult laryngoscopy scenario.
  Interventions: Device: tracheal tube

INTERVENTIONS:
Device: proceal laryngeal mask airway — In proceal laryngeal mask group, proceal laryngeal mask airway is inserted by novices.
  Other Names: LMA proceal
  Arms: proceal laryngeal mask airway
Device: tracheal tube — In tracheal tube group, tracheal tube is intubated by novices.
  Other Names: TaperGuard
  Arms: tracheal tube
Device: i-gel — In i-gel group, i-gel is inserted by novices.
  Arms: i-gel

SUMMARY:
The use of laryngeal mask airway or i-gel to manage airway may improve success rates, especially in difficult situations more than tracheal intubation.

DETAILED DESCRIPTION:
This study compares the insertion success rate and insertion time among the proceal laryngeal mask airway, i-gel, and tracheal tube. Following a short lecture, airway novices try to insert proceal laryngeal mask airway, i-gel, and tracheal tube into manikin with difficult laryngoscopy scenarios.

ELIGIBILITY:
Inclusion Criteria:

* medical student
* nurse
* no experience of insertion using tracheal tube, i-gel, and laryngeal mask airway

Exclusion Criteria:

* experience of insertion using tracheal tube, i-gel, and laryngeal mask airway

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the time of successful laryngeal mask, i-gel, or tracheal tube insertion attempt | intraoperative
  A blinded observer records the time of successful laryngeal mask, i-gel, or tracheal tube insertion attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Sangjin Park, M.D., Principal Investigator — Department of Anesthesiology and Pain Medicine, College of medicine, Yeungnam University, Daemyung-Dong, Nam-Gu, Daegu, Republic of Korea
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yeungnam University hospital, Daegu, South Korea